CLINICAL TRIAL: NCT01178697
Title: Three Injections of Intravitreal Bevasizumab Versus Two Injections of Intravitreal Triamcinolone in the Management of Branch Retinal Vein Occlusion
Brief Title: Intravitreal Bevasizumab Versus Intravitreal Triamcinolone in Central Retinal Vein Occlusion (CRVO)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Ophthalmic Research Center (Ambiguous)
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: 8886
Record Dates: First submitted 2010-08-02; First posted 2010-08-10 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-01

CONDITIONS: Central Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Intravitreal triamcinolone (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide
- Intravitreal bevasizumab (Active Comparator)
  Interventions: Drug: Bevasizumab

INTERVENTIONS:
Drug: Bevasizumab — Intravitreal, 1.25 mg, 3 times, one month apart.
  Arms: Intravitreal bevasizumab
Drug: Triamcinolone Acetonide — Intravitreal, 2 mg, 2 times, two months apart.
  Arms: Intravitreal triamcinolone

SUMMARY:
This randomized clinical trial is conducted to evaluate the effect of three intravitreal injections of bevasizumab versus two intravitreal injections of triamcinolone in acute central retinal vein occlusion. The outcomes are visual acuity and central macular thickness. The follow-up time is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Recent onset (less than 3 months) central retinal vein occlusion

Exclusion Criteria:

* Any previous intervention

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2010-01; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 6 months

SECONDARY OUTCOMES:
central macular thickness | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Hossein medical center, Tehran, Tehran Province, Iran